CLINICAL TRIAL: NCT07329387
Title: Electrophysiological Investigation of the Effectiveness of NMES Swallowing Difficulty Rehabilitation in Children With Cerebral Palsy
Brief Title: Effectiveness of NMES in Swallowing Rehabilitation in Children With CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Neslihan Altuntas Yilmaz, Principal Investigator, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/22
Record Dates: First submitted 2025-09-30; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Palsy (CP)
Keywords: Cerebral palsy; Dysphagia; Electric Stimulation Therapy; Suprahyoid muscle
MeSH Terms: conditions — Cerebral Palsy; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Study procedures The study was performed by a group of independent experts blinded to treatment allocation. The study was conducted by a group of independent experts blinded to the treatment allocation. An ear, nose, and throat specialist performed the physical examination, videofluoroscopic (Philips, Amsterdam, Netherlands) swallowing evaluation and electrophysiological evaluation. Unaware of the evaluation, swallowing rehabilitation was administered by a swallowing therapist. Subsequently, the patients were reevaluated by another ear, nose, and throat specialist using endoscopic assessment, unaware of the initial findings and observations. The randomization of patients was arranged by a 4th expert in physical medicine and rehabilitation. Experimental and control groups were formed. The patients completed the study without knowing which group they were assigned to. However, the swallowing therapist who administered the treatment was aware of the group assignments. Evalu
Who Masked: Outcomes Assessor
Masking Description: Randomization Randomization was performed in 32 patients according to the study criteria by independent (4nd) specialist. In accordance with the order of admission to the hospital, patients were randomly allocated by block randomization and a table of random numbers. The patients were numbered and grouped as 1.,4.,5.,8.,9.,… patients for Group 1, and 2.,3.,6.,7.,10.,... patients for Group 2. Allocation was performed before the initial evaluation. After randomization, 6 patients in Group 2 who were unable to adapt to rehabilitation programme were excluded and the study was completed with 26 patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMES (Experimental): In addition to the conventional swallowing rehabilitation approaches, neuromuscular electrical stimulation (NMES) was applied to the experimental group, while Sham-NMES was administered to the control group. For NMES applied to the suprahyoid muscle group, a frequency of 80 Hz with a pulse duration of 300-400 microseconds was used, and VitalStim therapy was administered for 40 minutes per session. In the Sham-NMES application, electrodes were placed on the same anatomical region, and the same amplitude and frequency settings were used as in the NMES protocol; however, no electrical current was delivered during the 40-minute session. To address ethical considerations, participants in the Sham-NMES group received 12 sessions of active NMES after completion of data collection, thereby minimizing potential bias.
  Interventions: Device: Neuromuscular Electrical Stimulation
- Sham-NMES (Sham Comparator): Sham NMES (Sham Neuromuscular Electrical Stimulation) is a placebo version of neuromuscular electrical stimulation used in clinical studies
  Interventions: Device: Sham Neuromuscular Electrical Stimulation

INTERVENTIONS:
Device: Neuromuscular Electrical Stimulation — For NMES applied to the suprahyoid muscle group, a 80 Hertz frequency, with a transition time of 300-400 microseconds, 40 minutes of Vital Stim application was performed
  Arms: NMES
Device: Sham Neuromuscular Electrical Stimulation — Sham NMES involves applying the electrical stimulation device without delivering therapeutic current, serving as a placebo control in randomized clinical trials
  Arms: Sham-NMES

SUMMARY:
Purpose: The aim is to investigate the effectiveness of NMES in the functional and electrophysiological rehabilitation of swallowing difficulties in dysphagic children with cerebral palsy.

Methods: Twenty-six children diagnosed with dysphagia, with a mean age of 7.02±2.40 years, were included in the study and randomly allocated into two groups (NMES,n=16;Sham NMES,n=10). In addition to swallowing rehabilitation, stimulation was applied to the groups. Participants were assessed using the Pediatric Eating Assessment Tool, Penetration-Aspiration Scale, Karaduman Chewing Performance Scale, Swallowing Ability and Function Evaluation and Electrophysiological Evaluation of the Suprahyoid Muscle in four consistencies.

DETAILED DESCRIPTION:
This study has already been completed; however, at the time of the study, registration in the public trial database had not been performed. Since the journal requires a registration number upon submission, we have completed a retrospective registration to fulfill this requirement. The registration reflects the actual study dates and ensures transparency and compliance with publication standard

ELIGIBILITY:
Inclusion Criteria:

* Patients whose relatives provided written informed consent
* Patients suitable for the planned intervention (assumed from context)

Exclusion Criteria:

* History of maxillary, head or neck surgery
* History of botulinum toxin treatment
* Structural oropharyngeal abnormality
* Gastroesophageal reflux disease (GERD)
* Receiving medical and/or physical therapy for dysphagia
* Severe cognitive, visual, auditory, or sensory impairments
* Drug use due to seizure or spasticity
* Serious pulmonary or cardiac disease
* Increased bleeding risk

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-01-02 (Actual)

PRIMARY OUTCOMES:
Pedi-EAT-10 | Baseline (pre-intervention)
  The Pedi-EAT-10 is a caregiver-administered, symptom-based questionnaire designed to screen for signs of oropharyngeal dysphagia in children aged 18 months and older. It consists of 10 items, each rated on a 5-point Likert scale (0 = no problem, 4 = severe problem), assessing observable feeding and swallowing difficulties.Time Frame: Baseline (pre-intervention)

OTHER OUTCOMES:
Pedi-EAT-10 | Baseline (pre-intervention) and immediately after the intervention.
  The Pedi-EAT-10 is a caregiver-administered, symptom-based questionnaire designed to screen for signs of oropharyngeal dysphagia in children aged 18 months and older. It consists of 10 items, each rated on a 5-point Likert scale (0 = no problem, 4 = severe problem), assessing observable feeding and swallowing difficulties.

CONTACTS AND LOCATIONS:
Locations (1):
- Nezahat Keleşoğlu Faculty of Health Sciences, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy and ethical concerns.